CLINICAL TRIAL: NCT01090752
Title: Effects of the PPAR-gamma Agonist Pioglitazone on Renal and Hormonal Responses to Salt in Diabetic and Hypertensive Subjects
Brief Title: Renal and Hormonal Effects of Pioglitazone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: University Hospital Geneva, University Hospital Geneva
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDAAA
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Results first posted 2010-04-08 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2009-01

CONDITIONS: Diabetes; Hypertension
Keywords: diabetes; blood pressure; pioglitazone; sodium; insulin resistance, renal function, sodium, pioglitazone
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Insulin Resistance | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Placebo Comparator): placebo-controlled, randomized, cross-over study
  Interventions: Drug: Pioglitazone; Drug: Metformin
- Metformine (Placebo Comparator): placebo-controlled, randomized, cross-over study was to explore the effects of pioglitazone (45 mg q.d. for 6 weeks) on the renal, hormonal and blood pressure responses to changes in sodium intake in a population prone to insulin resistance
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone — placebo-controlled, randomized, cross-over study was to explore the effects of pioglitazone (45 mg q.d. for 6 weeks) on the renal, hormonal and blood pressure responses to changes in sodium intake in a population prone to insulin resistance
  Other Names: Actos
  Arms: Pioglitazone
Drug: Metformin — placebo-controlled, randomized, cross-over study was to explore the effects of pioglitazone (45 mg q.d. for 6 weeks) on the renal, hormonal and blood pressure responses to changes in sodium intake in a population prone to insulin resistance
  Other Names: Glucophage; Glumetza; Fortamet; Riomet

SUMMARY:
This study examines the effects of pioglitazone on renal sodium handling in subjects prone to insulin resistance, i.e. diabetic and/or hypertensive subjects.

DETAILED DESCRIPTION:
Aim: Glitazones are powerful insulin sensitizers prescribed for the treatment of type 2 diabetes. Their use is however associated with fluid retention and an increased risk of congestive heart failure. We previously demonstrated that pioglitazone increases proximal sodium reabsorption in healthy volunteers. This study examines the effects of pioglitazone on renal sodium handling in subjects prone to insulin resistance, i.e. diabetic and/or hypertensive subjects.

Methods: In this double-blind, randomized, placebo-controlled, four-way, cross-over study, we examined the effects of pioglitazone (45mg daily during 6 weeks) or placebo on renal, systemic and hormonal responses to changes in sodium intake in 16 individuals, 8 with type 2 diabetic and 8 with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes
* Hypertension

Exclusion Criteria:

* Cardiac or renal diseases
* Anaemia
* Drugs like aspirin, non steroidal anti-inflammatory drugs and hormonal replacement therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Pechere-Bertschi, MD, Study Director — University Hospital, Geneva
Locations (1):
- Pechère-Bertschi Antoinette, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Zanchi A, Pechere-Bertschi A, Burnier M, Bonny O. Effects of pioglitazone on renal calcium excretion. J Clin Endocrinol Metab. 2011 Sep;96(9):E1482-5. doi: 10.1210/jc.2011-0373. Epub 2011 Jul 13. PMID 21752899
- [Derived] Zanchi A, Maillard M, Jornayvaz FR, Vinciguerra M, Deleaval P, Nussberger J, Burnier M, Pechere-Bertschi A. Effects of the peroxisome proliferator-activated receptor (PPAR)-gamma agonist pioglitazone on renal and hormonal responses to salt in diabetic and hypertensive individuals. Diabetologia. 2010 Aug;53(8):1568-75. doi: 10.1007/s00125-010-1756-2. Epub 2010 Apr 23. PMID 20414637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen subjects were examined, 8 with a diagnosis of type 2 diabetes (DM2) and 8 with a diagnosis of systemic hypertension (HTN). The participants were recruited by hospital placards detailing the study, and through ambulatory care centers in Lausanne and Geneva.
Pre-assignment Details: Each subject was randomised to receive either pioglitazone or placebo for 6 weeks, with a 2 week wash-out period between the two treatment phases. Randomisation of the sequences of placebo and active treatment periods were performed by a doctor having no contact with participants and clinicians.
Groups:
- Pioglitazone Low Salt/High Salt: a low salt and a high salt diet were given consequently and randomly during a week at the end of the pioglitazone phase
- Placebo Low Salt/High Salt: a low salt and a high salt diet were given consequently and randomly during a week at the end of the placebo phase
Period: Overall Study
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (2.8) | 52.5 (2.8) | 52.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Switzerland | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Effects of Pioglitazone on Renal Hemodynamics
Description: At the end of each treatment diet phase, renal clearances were performed for the determination of GFR and RBF
Time Frame: 2008
Measure: Mean (Standard Error); unit: ml/min/1.73m2
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt
Number analyzed (Participants) | 16 | 16
ml/min/1.73m2 | 68.0 (4.4) | 62.4 (5.0)

2. Primary Outcome: Effects of Pioglitazone on Sodium and Lithium Clearances
Description: At the end of each treatment and diet phase, 24 urine collections were collected for the determination of sodium and lithium clearances
Time Frame: 2007
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt
Number analyzed (Participants) | 16 | 16
ml/min | 1.05 (0.10) | 1.18 (0.13)

3. Primary Outcome: Effects of Pioglitazone on 24h Blood Pressure Control
Description: 24 hour blood pressure measurements were performed after each treatment/diet phase
Time Frame: march 2009
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt
Number analyzed (Participants) | 16 | 16
mmHg | 128 (5) | 129 (5)

4. Secondary Outcome: Effects of Pioglitazone on Salt Sensitivity
Time Frame: 2009
Reporting Status: Not Posted, anticipated posting 2010-06
Measure: Mean (Standard Error); unit: mmHg

ADVERSE EVENTS:
Arm/Group | Pioglitazone Low Salt/High Salt | Placebo Low Salt/High Salt
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The sample size may seem small but the cross over design of the study increased the statistical power. Each of 16 individuals was examined 4 times after the 4 different phases (pioglitazone-low salt, and high salt, placebo low salt and high salt).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No